CLINICAL TRIAL: NCT02659475
Title: Open-label Phentermine/Topiramate Extended Release (PHEN/TPM ER; Qsymia®) in Ten Subjects With Overweight or Obesity and DSM-V Binge Eating Disorder (BED)
Brief Title: Phentermine/Topiramate Extended Release in Binge Eating Disorder (BED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-2630
Record Dates: First submitted 2016-01-08; First posted 2016-01-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-01

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Qsymia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PHEN/TPM ER (Qsymia®) (Experimental): PHEN/TPM ER (Qsymia®)
  Interventions: Drug: PHEN/TPM ER (Qsymia®)

INTERVENTIONS:
Drug: PHEN/TPM ER (Qsymia®) — PHEN/TPM ER (Qsymia®)

SUMMARY:
The goal of this project is to evaluate the effectiveness and tolerability of the novel weight management medication PHEN/TPM ER (Qsymia®)along with nutritional and lifestyle modification counseling in the treatment of binge eating disorder (BED) in overweight or obese individuals.

DETAILED DESCRIPTION:
This is an exploratory open-label trial of PHEN/TPM ER (Qsymia®) in BED. It is hypothesized that PHEN/TPM ER (Qsymia®) will be an effective, safe, and well tolerated treatment for BED and propose to conduct a 1-site, 12-week, open-label, flexible dose study of PHEN/TPM ER (Qsymia®) in 10 outpatients, ages 18 through 65 years, with BED. It is also hypothesized that PHEN/TPM ER (Qsymia®) will reduce weight and binge eating behavior, and will be well tolerated. The primary objective is to show that PHEN/TPM ER (Qsymia®) along with nutritional and lifestyle modification counseling is effective in reducing weight in overweight or obese patients with BED. Secondary objectives are to show that PHEN/TPM ER (Qsymia®) is effective in reducing frequency of binge eating episodes and associated eating psychopathology and is safe and well tolerated in patients with BED.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ages of 18- 65 years, inclusive.
2. Subjects will meet DSM-5 criteria for a diagnosis of BED. These are:

   A. Recurrent episodes of binge eating. An episode of binge eating is characterized by both of the following:
   * Eating, in a discrete period of time (e.g., within a 2 hour period) an amount of food that is definitely larger than most people would eat in a similar period of time under similar conditions, and
   * Sense of lack of control over the eating (e.g., a feeling that one cannot stop eating or control what or how much one is eating)

   B. The binge eating episodes are associated with at least three of the following:
   * eating much more rapidly than normal
   * eating until uncomfortably full
   * eating large amounts of food when not feeling physically hungry
   * eating alone because of being embarrassed by how much one is eating
   * feeling disgusted with oneself, depressed, or feeling very guilty after overeating

   C. Marked distress regarding binge eating is present

   D. The binge eating occurs, on average, at least once a week for 3 months

   E. The binge eating is not associated with the recurrent use of inappropriate compensatory behavior as in bulimia nervosa and does not occur exclusively during the course of bulimia nervosa or anorexia nervosa
3. Subjects will be obese (defined as a BMI ≥ 30 mg/kg2) or overweight (defined as BMI ≥ 27 kg/m2 or greater) in the presence of at least one weight-related comorbidity, such as hypertension, type 2 diabetes mellitus, or dyslipidemia.
4. Subjects in treatment for a weight-related comorbidity (hypertension, type 2 diabetes mellitus, and/or dyslipidemia), must be on a stable medication regimen, defined as being on current dose of medication for at least 3 months prior to study enrollment.

Exclusion Criteria:

1. Current bulimia nervosa or anorexia nervosa.
2. Women who are pregnant, lactating, or of childbearing potential who are not using adequate contraceptive measures. The following are considered to be adequate methods of birth control: 1. Intrauterine device (IUD); 2. Barrier protection; 3. A contraceptive implantation system (Norplant); 4. Oral contraceptive pills; 5. A surgically sterile partner; and 6. Abstinence. Women who are >2years post-menopausal or surgically-sterile are not considered of childbearing potential. All female subjects will have a negative pregnancy test prior to randomization.
3. Subjects who are displaying clinically significant suicidality operationalized as a score ≥ 2 on item 9 of the Beck Depression Inventory (BDI) (21), or suicidal ideation on the Columbia-Suicide Severity Scale (C-SSRS) (22), or homicidality.
4. Subjects who are receiving a psychological (e.g., supportive psychotherapy, cognitive behavior therapy, interpersonal therapy) or weight loss (e.g., Weight Watchers) intervention for BED or weight management that was begun within the 3 months before study entry. Subjects who are receiving psychotherapy that was initiated prior to 3 months of the beginning of the study will be allowed to continue to receive their psychotherapy during the trial only if they agree to not make any changes in the frequency or nature of their psychotherapy during the course of the drug trial.
5. A DSM-5 diagnosis of a substance-related or addictive disorder (except a tobacco-related disorder) within the 6 months prior to enrollment.
6. A lifetime DSM-5 history of psychosis, mania or hypomania, or dementia.
7. History of any psychiatric disorder which might interfere with a diagnostic assessment, treatment, or compliance.
8. Clinically unstable medical disease, including cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease. Subjects should be biochemically euthyroid to enter the study.
9. Have a history of a structural cardiac abnormality, valvular cardiac disease, cardiomyopathy, serious heart rhythm abnormality, coronary artery disease, stroke, or other serious cardiovascular problem.
10. History of seizure disorder, including clinically-significant febrile seizures in childhood.
11. Subjects with glaucoma or hyperthyroidism.
12. Have an ECG with significant arrhythmias or conduction abnormalities, which in the opinion of the physician investigator preclude study participation.
13. Have clinically relevant abnormal laboratory results.
14. Subjects requiring treatment with any drug which might interact adversely with or obscure the action of the study medication. This includes anti-obesity drugs, psychostimulants, wake-promoting agents, drugs with serotonergic properties, antidepressants, and antipsychotics.
15. Subjects who have received any psychotropic medications (other than hypnotics) within four weeks prior to randomization, including monoamine oxidase inhibitors, tricyclics, selective serotonin reuptake inhibitors, antipsychotics, mood stabilizers, or psychostimulants.
16. Subjects who have received investigational medications or depot neuroleptics within three months prior to randomization.
17. Subjects who have a known allergy to PHEN/TPM ER (Qsymia®) or its constituents.
18. Subjects with a urine drug screen positive for a drug that, in the opinion of the investigator, is being abused.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
change in weight | from baseline visit (week 0) to final visit or early termination
  Weight will be measured at all study visits - screen, baseline (week 0), and weeks 2, 4, 6, 8, 10. 12

CONTACTS AND LOCATIONS:
Overall Officials: Anna Guerdjikova, PhD,LISW, Principal Investigator — Lindner Center of HOPE
Locations (1):
- Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Derived] Guerdjikova AI, Williams S, Blom TJ, Mori N, McElroy SL. Combination Phentermine-Topiramate Extended Release for the Treatment of Binge Eating Disorder: An Open-Label, Prospective Study. Innov Clin Neurosci. 2018 Jun 1;15(5-6):17-21. PMID 30013815